CLINICAL TRIAL: NCT03437200
Title: Phase II Trial in Inoperable œsophageal Cancer Evaluating the Feasibility of the Combination of Definitive Chemoradiation With the Immune Checkpoint Blockers Nivolumab +/- Ipilimumab
Brief Title: Combination of Chemoradiation With Immunotherapy in Inoperable œsophageal Cancer
Acronym: CRUCIAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1714; 2018-000053-53 (EudraCT Number)
Record Dates: First submitted 2018-02-06; First posted 2018-02-19 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Inoperable œsophageal Cancer
Keywords: œsophageal cancer nivolumab ipilimumab
MeSH Terms: interventions — Nivolumab; Ipilimumab; Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Chemoradiation + Nivolumab (Experimental): All patients will receive standard fractionation radiation therapy (RT) scheme: 50Gy in 25 fractions over 5 weeks (i.e. 2Gy per fraction), concurrently with 3 cycles of 2 weeks of FOLFOX followed by 3 cycles of 2 weeks of FOLFOX without RT.
  Induction phase: Nivolumab IV 240 mg on days 1, 15 and 29 followed by a maintenance phase (to start on day 43) of Nivolumab IV 240 mg q2 weekly for up to 1 year.
  Interventions: Drug: Nivolumab; Other: Chemoradiation
- Arm B: Chemoradiation + Nivolumab + Ipilimumab (Experimental): Same as arm A + induction phase: Ipilimumab IV 1 mg/kg on day 1 followed by a maintenance phase (to start on day 43) of Ipilimumab IV 1 mg/kg q6 weekly for up to 1 year
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Other: Chemoradiation

INTERVENTIONS:
Drug: Nivolumab — Induction phase: Nivolumab IV 240 mg on days 1, 15 and 29 followed by a maintenance phase (to start on day 43) of Nivolumab IV 240 mg q2 weekly for up to 1 year.
Drug: Ipilimumab — Induction phase: Ipilimumab IV 1 mg/kg on day 1 followed by a maintenance phase (to start on day 43) of Ipilimumab IV 1 mg/kg q6 weekly for up to 1 year.
  Arms: Arm B: Chemoradiation + Nivolumab + Ipilimumab
Other: Chemoradiation — All patients will receive standard fractionation radiation therapy (RT) scheme: 50Gy in 25 fractions over 5 weeks (i.e. 2Gy per fraction), concurrently with 3 cycles of 2 weeks of FOLFOX (oxaliplatin 85 mg/m2, leucovorin 200 mg/m2, bolus fluorouracil 400 mg/m2, and infusional fluorouracil 1600 mg/m2 over 48 h), followed by 3 cycles of 2 weeks of FOLFOX without RT.

SUMMARY:
The main objective of the trial is to assess the feasibility and the safety of the addition of immunotherapy with PD-1 antibody nivolumab +/- CTLA-4 antibody ipilimumab to concomitant chemoradiation therapy (CRT) in inoperable patients with early or locally advanced oesophageal cancer and to select the more promising experimental arm among the two possible combinations in terms of activity (based on progression free survival (PFS) at 12 months according to RECIST 1.1) for further evaluation in a phase III trial.

The secondary objectives will aim to evaluate progression-free survival, failure-free survival and overall survival and pattern of progression (including incidence of distance metastasis).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven oesophageal squamous cell carcinoma or adenocarcinoma
* Both early stage and locally advanced tumor patients (according to TNM staging version 8):
* T1, N1-3, M0 after complete work-up
* T2, N0-3, M0 after complete work-up
* T3, N0-3, M0
* Patient eligible for definitive chemoradiation and not considered for primary surgery after multidisciplinary meeting decision or patient refuses to undergo surgery
* Subject must be previously untreated with systemic treatment given as primary therapy for advanced or metastatic disease
* At least one measurable lesion by CT scan or MRI based on RECIST version 1.1 with radiographic tumor assessment performed within 28 days prior to randomization
* Availability of adequate tissue in terms of quality and quantity for immunohistochemical staining for PDL-1
* WHO performance status 0 or 1
* Adequate organ function within 14 days prior to randomization

Exclusion Criteria:

* Cancer of cervical oesophagus (15 to 19 cm from dental ridge)
* Known Her2 positive adenocarcinoma
* Weight loss > 15 % over the last 3 months without improvement after nutritional support
* Patient with cardiac dysfunction e.g. symptomatic congestive heart failure, uncontrolled hypertension
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS), hepatitis B or hepatitis C.
* Any prior treatment for advanced disease including treatment with an anti-Programmed Death receptor-1 (PD-1), anti-Programmed Death-1 ligand-1 (PD-L1), anti-PD-L2, anti-cytotoxic T lymphocyte associated antigen-4 (anti-CTLA-4) antibody or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Live vaccines within 30 days prior to the first dose of study therapy. Examples of live vaccines include, but are not limited to the following: measles, mumps, rubella, chicken pox, yellow fever, H1N1 flu, rabies, BCG, and typhoid vaccine
* History of hypersensitivity to study drugs or any excipient (refer to SmPCs for ipilimumab, nivolumab, 5-FU and oxaliplatin)
* Current participation or treatment with an investigational agent or use of an investigational agent within 4 weeks of the first dose of study treatment
* Serious comorbidity or life expectancy less than one year
* Contraindication to chemoradiation therapy
* Treatment history of radiotherapy
* Child-Pugh B/C and patients with history of acute or chronic pancreatitis
* Patient with Type I diabetes mellitus, or skin disorders
* Known severe systemic autoimmune disease affecting the lungs or the bowel
* Known contraindication to CT scans with IV contrast
* Chronic use of immunosuppressive agents and/or systemic corticosteroids or any use in the last 15 days prior to enrollment
* Active autoimmune disease that has required systemic treatment in past 2 years
* Autoimmune paraneoplastic syndrome requiring immunosuppressive or dedicated treatment
* History of any other hematologic or primary solid tumor malignancy, unless in remission for at least 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
12-Month Progression-free survival using RECIST 1.1 | 3.8 years from first patient in
  The analysis of the 12-Month Progression-free survival rate (PFS-12) will be done when all patients achieved at least 15 months follow-up (12 months for the primary endpoint plus 100 days after the end of the protocol treatment).

SECONDARY OUTCOMES:
Best overall response according to RECIST 1.1 | 3.8 years from first patient in
Pattern of first cause of progression (either local relapse/progression,either regional relapse/progression, either distant metastasis) | 3.8 years from first patient in
Progression-free survival using RECIST 1.1 | 3.8 years from first patient in
Failure-free survival | 3.8 years from first patient in
Overall survival | 3.8 years from first patient in
Percentage of patients receiving the planned chemoradiation | 3.8 years from first patient in
Relative dose intensity of oxaliplatinum | 3.8 years from first patient in
  The dose intensity and relative dose intensity of treatments will be presented by drug and by treatment arm using median, range and interquartile range.
Relative dose intensity of 5FU | 3.8 years from first patient in
  The dose intensity and relative dose intensity of treatments will be presented by drug and by treatment arm using median, range and interquartile range.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Deutsch, Principal Investigator — INSTITUT GUSTAVE ROUSSY, Paris, France; Markus Moehler, Principal Investigator — UNIVERSITY MEDICAL CENTER MAINZ, Germany
Locations (7):
- France (2):
  - Assistance Publique - Hopitaux de Paris - La Pitie Salpetriere, Paris
  - Institut Gustave Roussy, Villejuif
- Spain (5):
  - Hospital Del Mar, Barcelona
  - Institut Catala d'Oncologia - ICO Badalona - Hospital De Mataro, Barcelona
  - Institut Catala d'Oncologia - ICO L'Hospitalet - Hospital Duran i Reynals (Institut Catala D'Oncologia), Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario 12 De Octubre, Madrid